CLINICAL TRIAL: NCT02635906
Title: Effectiveness of Reduced in Bed Rest After Coronary Arteriography or Coronary Angioplasty in Patients With Acute Coronary Syndrome: 4 Hours Versus 2 h.Clinical Trial
Brief Title: Reduced in Bed Rest After Coronary Arteriography or Coronary Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Vinicius Batista Santos, Nursing Coordinator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 49068315.0.0000.5505
Record Dates: First submitted 2015-11-30; First posted 2015-12-21 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Acute Coronary Syndrome
Keywords: BED REST; CORONARY ANGIOPLASTY
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 hours (Experimental): after coronary arteriography or coronary angioplasty, will be removal the introducer and the patient will be in bed rest for two hours
  Interventions: Other: 2 hours
- 4 hours (Active Comparator): after coronary arteriography or coronary angioplasty, will be removal the introducer and the patient will be in bed rest for four hours
  Interventions: Other: 4 hours

INTERVENTIONS:
Other: 2 hours — BED REST FOR TWO HOURS AFTER CORONARY ARTERIOGRAPHY OR CORONARY ANGIOPLASTY
  Other Names: reduced bed rest
  Arms: 2 hours
Other: 4 hours — BED REST FOR FOUR HOURS AFTER CORONARY ARTERIOGRAPHY OR CORONARY ANGIOPLASTY
  Other Names: four hours group
  Arms: 4 hours

SUMMARY:
This is a randomized clinical trial with a control group, based on the guidelines of the CONSORT 2010. The interventional group will be in a bed rest for two hours after introducer removal in patients submitted a coronary arteriography or coronary angioplasty and the control group will follow the standard nursing care for four hours.

DETAILED DESCRIPTION:
This is a randomized clinical trial with a control group, based on the guidelines of the CONSORT 2010. It will be held in the cardiology unit of a public hospital in the city of São Paulo in patients admitted with Acute Coronary Syndrome undergoing coronary arteriography or coronary angioplasty by femoral arterial. Patients with hemodynamic instability will be excluded before and after the ATC, patients using oral anticoagulants presenting INR greater than 2; patients using inhibitors IIB / IIIa; patients with history of blood dyscrasias; patients undergoing invasive procedure again less than 24 hours; patients with previous diagnosis of arterial insufficiency and patients at the time of withdrawal of the introducer presenting systolic blood pressure greater than 180 mmHg and diastolic than 100 mmHg. After removing the introducer the interventional group will be in a bed rest for two hours and the control group will follow the standard nursing care for four hours. Will be assessed the following indicators: bruising, bleeding, pedis pulse and popliteal, presence of blast at the puncture site after removal of the introducer, peripheral perfusion, presence of pulsatile mass, back pain, low back pain, paresthesias, urinary retention, muscle aches, use of painkillers and erythrocyte level.

These indicators will be assessed prior to the procedure, immediately after removing the introducer, 6 hours after the removal of the introducer, 12 hours after removal of the introducer and 24 hours after removal of the introducer. Vascular outcomes will be considered the appearance of bruising, bleeding, pseudoaneurysm, arteriovenous fistula, retroperitoneal hematoma and acute arterial occlusion. Related to patient outcomes will be considered the complaints back pain, back pain, muscle pain, paresthesia and urinary retention. The assessment team will be composed of three nurses specialists in cardiology with a minimum of one year experience in patient care after the ATC. For this study will be presented by the principal investigator to the patient the study objectives, possible risks and complications and the study protocol, and if the patient agrees to participate in it will be delivered the Statement of Consent. The collected data regarding the patients included in the survey will be entered initially in a Microsoft Excel® 2010 software and later transferred to an electronic database software SPSS (Statistical Package for Social Sciences) version 20.0 and, then submitted to descriptive statistical analysis and comparison analysis between groups.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted with Acute Coronary Syndrome undergoing coronary arteriography or coronary angioplasty by femoral arterial.

Exclusion Criteria:

* patients with hemodynamic instability will be excluded before and after the ATC,
* patients using oral anticoagulants presenting INR greater than 2;
* patients using inhibitors IIB / IIIa;
* patients with history of blood dyscrasias;
* patients undergoing invasive procedure again less than 24 hours;
* patients with previous diagnosis of arterial insufficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Back Pain, Lumber Pain and Muscle Pain | 1 hour after the bed rest
  This outcome will be measured in relation to presence or absence. The presence and will Assess by means of a visual analog scale of 0 to 10, whereas the smallest value as no pain and the largest value as unbearable pain.

SECONDARY OUTCOMES:
Haematoma | 24 hours after the coronary angioplasty
  This outcome will be measured in relation to presence or absence. The presence and will measured with a millimeter ruler taking.
Bleeding | 24 hours after the coronary angioplasty
  This outcome will be measured when appear blood in a bandage or when the haemoglobin decrease more than 3g/d.
Pseudoaneurysm, Arteriovenous Fistula: Retroperitoneal hematoma, Acute Arterial Occlusion: | 24 hours after the coronary angioplasty
  This outcome will be measured in relation to presence or absence by ultrasound.
Urinary retention, Paresthesia | 1 hour after the bed rest
  This outcome will be measured in relation to presence or absence.

CONTACTS AND LOCATIONS:
Overall Officials: VINICIUS B SANTOS, MASTER, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital São Paulo - Cardiology Unit, São Paulo, Brazil